CLINICAL TRIAL: NCT04230746
Title: Effect of Antibiotics on Urinary Microbiome: Randomized Trial
Brief Title: Effect of Antibiotics on Urinary Microbiome
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: funding , recruitment issues
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00224835
Record Dates: First submitted 2019-12-27; First posted 2020-01-18 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Microtia; UTI; Bacteriuria; Antibiotic Resistant Infection; Antibiotics Causing Adverse Effects in Therapeutic Use
Keywords: microbiome; antibiotics; resistance; flora
MeSH Terms: conditions — Congenital Microtia; Bacteriuria | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: Planning to study the urine microbiota at baseline and after administration of bactrim antibiotics in healthy volunteers. Will intermittently collect voided urine specimens for 16 s DNA analysis over a period of 6 months after 2 weeks of bactrim or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Drug will be blinded to all.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants will be recruited and enrolled. Participants will be surveyed regarding environmental, health, and behavioral practices. (Instrument 1) . Then a clean catch urine specimen will be collected. Participants will be provided with placebo to be taken twice daily. This will be considered day 0. Participants will then be instructed to take the study drug twice daily and return on Day 2, Day 5, Day 10, Day 30, and Day 180 for additional clean-catch urine specimen.
  Interventions: Drug: Placebo oral tablet
- Bactrim (Experimental): Participants will be recruited and enrolled. Participants will be surveyed regarding environmental, health, and behavioral practices. (Instrument 1) . Then a clean catch urine specimen will be collected. Participants will be provided with Bactrim 800/120 to take twice daily. This will be considered day 0. Participants will then be instructed to take the study drug twice daily and return on Day 2, Day 5, Day 10, Day 30, and Day 180 for additional clean-catch urine specimen.
  Interventions: Drug: Bactrim DS 800Mg-160Mg Tablet

INTERVENTIONS:
Drug: Bactrim DS 800Mg-160Mg Tablet — To study effect on urinary microbiome
  Other Names: bactrim, trimethoprim sulfamethoxazole, Septra, sulfatrim
  Arms: Bactrim
Drug: Placebo oral tablet — To study effect on urinary microbiome
  Arms: Placebo

SUMMARY:
Planning to study urine microbiota at baseline and after administration of bactrim antibiotics in healthy volunteers. Will intermittently collect voided urine specimens for 16 s DNA analysis over a period of 6 months after 2 weeks of bactrim or placebo.

DETAILED DESCRIPTION:
Urinary tract infections (UTI) are the most common type of human bacterial disease, prompting more than 10 million physician office visits annually at a healthcare cost of over $1 billion dollars. Treatment of UTI is typically empiric or culture-driven antibiotics which are associated with ever increasing bacterial resistance. Over the last decade, The Human Microbiome Project has established that even 'culture-negative' urine represents a diverse ecosystem of bacteria. Despite broad use of antibiotics to cure disease for the past 90 years, the broader impact of antibiotics on typical flora are not well understood. Antibiotics are also commonly used as prophylaxis for surgical procedures in the urinary tract altering patient outcomes in unforeseen ways. Despite widespread utilization of antibiotics, the longitudinal impact on the dynamic intravesical environment remains completely unknown.

Dysbiosis in the microbiome has been suggested as a causative agent in a wide range of disease: arthritis, metabolic disorders, neurologic disease, inflammatory bowel conditions, and cancer. Yet there remains a fundamental knowledge gap regarding the short and long-term effect of antibiotics on microbiota communities. Specifically within the urinary tract, variance in baseline commensal organisms have been associated with interstitial cystitis, overactive bladder, frequent symptomatic urinary tract infection and potentially cancer development. The study of microbiota reveal pathways and mechanisms that play important roles in immunological response and health but studies typically are limited to the gut.

To address this knowledge gap, the investigators plan a placebo controlled randomized trial to test the longitudinal impact of 10 days of trimethoprim-sulfamethoxazole on the urinary microbiome in healthy adults. Data collection for individual participants will persist for a period of 6 months. The investigators hypothesize antibiotic administration contributes to a rise in bacterial resistance and directly leads to urine microbiome dysbiosis. The investigators further hypothesize the urinary microbiome does not return to baseline, with loss of certain bacteria permanent during the study period. While the investigators' study is groundbreaking and novel, the feasibility of the investigators' experimental plan has been previously demonstrated in the study of the salivary and gut microbiome. Ultimately the investigators anticipate even a single course of antibiotic treatment may increase the risk of bacterial resistance and lead to long-lasting shifts in the urinary microbiome. If confirmed, this knowledge will directly influence clinical decision making in antibiotic selection, duration, and utility.

ELIGIBILITY:
Exclusion Criteria:

* Diagnosed or suspected urinary tract infection in prior 6 months
* Treated with antibiotics for any reason in prior 6 months
* Allergy to sulfa
* Under 18
* Pregnant or planning to become pregnant in the next 12 months by self report (as is the clinical standard for prescribing this medication for suspected or proven UTI treatment)
* Use indwelling or intermittent urinary hardware or implant such as supra-pubic tube or catheter
* Neurogenic bladder
* Baseline renal insufficiency
* Glucose-6-phosphate dehydrogenase deficiency
* Taking angiotensin converting enzyme
* Angiotensin receptor blocker
* Nursing
* HIV/AIDS
* On Immunosuppressant drugs
* On Chemotherapy/Immunotherapy
* Liver dysfunction
* On the following medications: DOFETILIDE, METHENAMINE & LEVOMETHADYL; WARFARIN & Methotrexate; GEMIFLOXACIN, DIGOXIN, PYRIMETHAMINE, CLASS IA ANTIARRHYTHMIC AGENTS (Quinidine, procainamide, disopyramide), TRICYCLIC ANTIDEPRESSANTS (amitriptyline, desipramine, doxepin, Imipramine, nortriptyline, amoxapine, clomipramine, maprotiline, trimipramine, and protriptyline), LEUCOVORIN CALCIUM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Microbiome flora number of organisms | At Baseline, Day 2, Day 5, Day 10, Day 30, and Day 180 of study
  Analysis of 16S rRNA gene amplicon data to determine number of varied organisms (genus and species).
Change in Microbiome flora percentage distribution of organisms | At Baseline, Day 2, Day 5, Day 10, Day 30, and Day 180 of study
  Analysis of 16S rRNA gene amplicon data to determine the percent distribution of organisms (microbiologic genus and species).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Cohen, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No